CLINICAL TRIAL: NCT00026871
Title: Clinical Evaluation of a Laser Heated, Fiberoptic-Coupled Radiation Dose Verification System
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 970129; 97-C-0129
Record Dates: First submitted 2001-11-14; First posted 2001-11-15 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-05

CONDITIONS: Neoplasm
Keywords: Non-Therapeutic; Radiation Therapy; Dosimetry; Dose-Rate; Fiberoptic
MeSH Terms: conditions — Neoplasms | interventions — Radiotherapy

INTERVENTIONS:
Procedure: Radiotherapy

SUMMARY:
We propose to determine the response of a newly developed laser heated, vycor glass fiberoptic radiation dosimetry system to ionizing radiation in a clinical radiotherapy environment. Present systems measure only total dose or have limitations, such as instability, non-linearity, excessive size or a decoupled measurement system, making them unsuitable in a variety of clinical applications. This fiberoptic coupled dosimetry system is a new and innovative technology application which allows on-line measurement of instantaneous dose rate and total dose never before achievable. It offers a clear advantage in patient treatment delivery, allowing on-line corrections essential to a new generation of radiotherapy treatment machines with development of beam intensity modulation as an adjunct to 3D conformal therapy. It also has the advantage of submillimeter size and is minimally invasive, making it ideal for brachytherapy.

This system has the potential for stable, accurate, reproducible, clinically feasible measurements of total dose and dose rate. The output of this system will be measured under various clinical conditions encountered in a clinical setting and compared against existing thermolumeniscent and diode dosimetry standards. Initial measurements will use a tissue equivalent phantom for depth dose and accuracy measurements. Additional studies will include dosimetric measurements of routine clinical treatment setups on patients receiving therapeutic irradiation.

DETAILED DESCRIPTION:
We propose to determine the response of a newly developed laser heated, vycor glass fiberoptic radiation dosimetry system to ionizing radiation in a clinical radiotherapy environment. Present systems measure only total dose or have limitations, such as instability, non-linearity, excessive size or a decoupled measurement system, making them unsuitable in a variety of clinical applications. This fiberoptic coupled dosimetry system is a new and innovative technology application which allows on-line measurement of instantaneous dose rate and total dose never before achievable. It offers a clear advantage in patient treatment delivery, allowing on-line corrections essential to a new generation of radiotherapy treatment machines with development of beam intensity modulation as an adjunct to 3D conformal therapy. It also has the advantage of submillimeter size and is minimally invasive, making it ideal for brachytherapy.

This system has the potential for stable, accurate, reproducible, clinically feasible measurements of total dose and dose rate. The output of this system will be measured under various clinical conditions encountered in a clinical setting and compared against existing thermolumeniscent and diode dosimetry standards. Initial measurements will use a tissue equivalent phantom for depth dose and accuracy measurements. Additional studies will include dosimetric measurements of routine clinical treatment setups on patients receiving therapeutic irradiation.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients receiving either external beam radiotherapy or a radioactive implant under established primary clinical protocols at the NCI or the National Naval Medical Center.

Patients must be willing to have the additional measurements performed and sign an informed consent.

EXCLUSION CRITERIA:

Pediatric and cognitively impaired subjects will not be eligible for this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 1997-07; Study Completion 2006-05

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States